CLINICAL TRIAL: NCT03436615
Title: A Phase 2 Multi-Center, Randomized, Double-Blind, Vehicle-Controlled Ascending Dose Study of SB206 in Subjects With Molluscum Contagiosum
Brief Title: A Study to Evaluate the Safety and Efficacy of SB206 in Subjects With Molluscum Contagiosum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NI-MC201
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Molluscum Contagiosum
MeSH Terms: conditions — Molluscum Contagiosum | interventions — berdazimer sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SB206 4% (Experimental): SB206 4% topically twice daily
  Interventions: Drug: SB206 4%
- SB206 8% (Experimental): SB206 8% topically twice daily
  Interventions: Drug: SB206 8%
- SB206 12% (Experimental): SB206 12% topically once or twice daily
  Interventions: Drug: SB206 12%
- Placebo (vehicle gel) (Placebo Comparator): Vehicle Gel topically once or twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB206 4% — Twice daily
  Other Names: NVN1000
  Arms: SB206 4%
Drug: SB206 8% — Twice daily
  Other Names: NVN1000
  Arms: SB206 8%
Drug: SB206 12% — Once or twice daily
  Other Names: NVN1000
  Arms: SB206 12%
Drug: Placebo — Once or twice daily
  Other Names: Vehicle Gel
  Arms: Placebo (vehicle gel)

SUMMARY:
This is a phase 2 multi-center, randomized, double-blind, vehicle-controlled ascending dose study to be conducted in non-immunocompromised subjects with molluscum contagiosum.

DETAILED DESCRIPTION:
This is a phase 2 multi-center, randomized, double-blind, vehicle-controlled ascending dose study to be conducted in up to approximately 192 or 256 non-immunocompromised subjects with molluscum contagiosum. Subjects who satisfy entry criteria will be randomized 3:1 to ascending, sequential dose cohorts of SB206. The highest tolerated dose will also be run in a cohort once daily. Approximately 64 subjects will be randomized to each cohort. Subjects will be treated once daily, twice daily or three times a week for up to 12 weeks. After 30 subjects randomized in a cohort have completed 2 weeks of treatment, the Data Safety Monitoring Board (DSMB) will review the available unblinded safety and tolerability data. The DSMB will determine if the data supports escalating to the next highest dose for the next cohort or if the data shows the dose is not tolerable decreasing to the next lower dose or frequency for the next cohort.

ELIGIBILITY:
Inclusion Criteria:

* Be 2 years of age or older, and in good general health;
* Have signed written informed consent form by a parent or legal guardian (assent form where required);
* Have between 3 and 70 MC at baseline, excluding periocular (within 2 cm circumference of the eye) and lesions on the labia and penis;
* Females 10 years of age and older must have a negative urine pregnancy test prior to randomization;
* Females 10 years of age and older must agree to use an effective method of birth control during the course of the study and for 30 days after their final study visit;
* Be willing and able to follow study instructions and likely to complete all study requirements.

Exclusion Criteria:

* Are immunosuppressed, have immunodeficiency disorder, or are on immunosuppressive treatment;
* Have agminated MC that could make it difficult to provide accurate lesion counts;
* Have active atopic dermatitis with intense erythema and/or excoriations, that impact currently or could impact at any point during the study the ability to count MC lesions;
* Have significant eczematous reactions or other skin disease surrounding MC that may impact the ability to count lesions;
* Have received treatment with topical calcineurin inhibitors or steroids on MC or within 2 cm of MC lesions within 14 days prior to baseline;
* Have received treatment for MC during the 14 days prior to baseline with podophyllotoxin, imiquimod, cantharidin, sinecatechins, topical retinoids, oral or topical zinc, or other homeopathic or OTC products including, but not limited to, Zymaderm and tea tree oil, cimetidine and other histamine H2 receptor antagonists;
* Have received surgical procedures (cryotherapy, curettage, other) within 28 days prior to baseline;
* Have MC only in periocular area;
* Have MC only on the labia or penis;
* Female subjects who are pregnant, planning a pregnancy or breastfeeding;
* Have confirmed methemoglobin level of >3.0% at Baseline using a pulse co-oximeter;
* Have know hypersensitivity to any ingredients of SB206 or Vehicle Gel including excipients;
* Have participated in a previous study with NVN1000;
* Have participated in any other trial of an interventional investigational drug or device within 30 days or concurrent participation in another interventional research study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-11-03 (Actual); Study Completion 2018-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Maeda-Chubachi, MD, Study Chair — Novan, Inc.
Locations (18):
- United States (18):
  - Premier Site# 266, Scottsdale, Arizona
  - Premier Site# 260, Santa Ana, California
  - Premier Site# 257, Thornton, Colorado
  - Premier Site# 264, Doral, Florida
  - Premier Site# 116, Newnan, Georgia
  - Premier Site# 251, Indianapolis, Indiana
  - Premier Site# 253, Lenexa, Kansas
  - Premier Site# 117, Louisville, Kentucky
  - Premier Site# 182, Las Vegas, Nevada
  - Premier Site# 252, Norman, Oklahoma
  - Premier Site# 237, Gresham, Oregon
  - Premier Site# 259, Charleston, South Carolina
  - Premier Site# 255, Mt. Pleasant, South Carolina
  - Premier Site# 131, Houston, Texas
  - Premier Site# 167, Houston, Texas
  - Premier Site# 224, San Antonio, Texas
  - Premier Site# 256, Salt Lake City, Utah
  - Premier Site# 267, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: SB206 4% BID: SB206 4% topically twice daily
- Cohort 2: SB206 8% BID: SB206 8% topically twice daily
- Cohort 3: SB206 12% BID: SB206 12% topically twice daily
- Cohort 4: SB206 12% QD: SB206 12% topically once daily
Period: Overall Study
Arm/Group | Cohort 1: SB206 4% BID | Cohort 2: SB206 8% BID | Cohort 3: SB206 12% BID | Cohort 4: SB206 12% QD | Placebo (Vehicle Gel)
Started | 47 | 48 | 47 | 48 | 66
Completed | 38 | 40 | 39 | 43 | 61
Not Completed | 9 | 8 | 8 | 5 | 5

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: SB206 4% BID | Cohort 2: SB206 8% BID | Cohort 3: SB206 12% BID | Cohort 4: SB206 12% QD | Placebo (Vehicle Gel) | Total
Number analyzed (Participants) | 47 | 48 | 47 | 48 | 66 | 256
Age, Customized [Count of Participants; unit: Participants]
  ≥2 years of age | 47 | 48 | 47 | 48 | 66 | 256
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 22 | 25 | 27 | 123
  Male | 25 | 21 | 25 | 23 | 39 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 11 | 16 | 8 | 15 | 56
  Not Hispanic or Latino | 41 | 37 | 31 | 40 | 51 | 200
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 0 | 2
  Asian | 2 | 1 | 1 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 3 | 0 | 2 | 1 | 7
  White | 40 | 42 | 44 | 44 | 58 | 228
  More than one race | 3 | 1 | 0 | 1 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 48 | 47 | 48 | 66 | 256
Baseline number of Molluscum lesions [Mean (Standard Deviation); unit: Molluscum lesions] — Population: It was pre-planned to analyze the SB206 Arms/Groups and the Placebo Arm/Group separately.
  Molluscum lesions
    SB206: number analyzed (Participants) | 47 | 48 | 47 | 48 | 0 | 190
    SB206 | 21.7 (17.23) | 19.0 (14.37) | 18.8 (16.15) | 17.6 (16.55) |  | 19.3 (16.05)
    Placebo (vehicle gel): number analyzed (Participants) | 0 | 0 | 0 | 0 | 66 | 66
    Placebo (vehicle gel) |  |  |  |  | 18.3 (14.47) | 18.3 (14.47)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Complete Clearance at Week 12
Description: Percent (proportion) of subjects with complete clearance of all treatable MC at Week 12. This was measured by dividing the number of subjects who showed complete clearance by the number in that treatment group (this represents our primary outcome variable).
Time Frame: 12 weeks
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SB206 4% BID | Cohort 2: SB206 8% BID | Cohort 3: SB206 12% BID | Cohort 4: SB206 12% QD | Placebo (Vehicle Gel)
Number analyzed (Participants) | 38 | 39 | 37 | 43 | 60
Participants | 5 | 16 | 13 | 18 | 12

2. Secondary Outcome: Proportion of Subjects Achieving Complete Clearance at Each Visit
Description: Proportion of subjects achieving complete clearance of all treated molluscum contagiosum lesions at each visit.
Time Frame: Week 1; Week 2; Week 4; Week 8; Week 12
Population: mITT population
Measure: Number; unit: participants
Arm/Group | Cohort 1: SB206 4% BID | Cohort 2: SB206 8% BID | Cohort 3: SB206 12% BID | Cohort 4: SB206 12% QD | Placebo (Vehicle Gel)
Number analyzed (Participants) | 38 | 39 | 37 | 43 | 60
participants
  Week 1 proportion of subjects achieving complete clearance.: number analyzed (Participants) | 35 | 37 | 36 | 43 | 57
  Week 1 proportion of subjects achieving complete clearance. | 0 | 1 | 0 | 1 | 0
  Week 2 proportion of subjects achieving complete clearance.: number analyzed (Participants) | 38 | 39 | 36 | 42 | 59
  Week 2 proportion of subjects achieving complete clearance. | 1 | 1 | 1 | 3 | 1
  Week 4 proportion of subjects achieving complete clearance.: number analyzed (Participants) | 37 | 39 | 36 | 41 | 59
  Week 4 proportion of subjects achieving complete clearance. | 1 | 3 | 3 | 5 | 2
  Week 8 proportion of subjects achieving complete clearance.: number analyzed (Participants) | 37 | 37 | 36 | 41 | 58
  Week 8 proportion of subjects achieving complete clearance. | 3 | 7 | 10 | 11 | 6
  Week 12 proportion of subjects achieving complete clearance.: number analyzed (Participants) | 34 | 39 | 36 | 43 | 59
  Week 12 proportion of subjects achieving complete clearance. | 5 | 16 | 13 | 18 | 12

3. Secondary Outcome: Time to First Complete Clearance
Description: Median time to reach first complete clearance of all molluscum contagiosum lesions (Kaplan-Meier estimate)
Time Frame: Week 12
Population: mITT
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 1: SB206 4% BID | Cohort 2: SB206 8% BID | Cohort 3: SB206 12% BID | Cohort 4: SB206 12% QD | Placebo (Vehicle Gel)
Number analyzed (Participants) | 38 | 39 | 37 | 43 | 60
Days | NA [13 to 85] — This was a Kaplan-Meier estimate and the median wasn't reached in the SB206 4% BID cohort due to insufficient numbers of participants achieving complete clearance. | 100.0 [11 to 100] | 91.0 [16 to 91] | 85.0 [8 to 86] | 93.0 [17 to 93]

4. Secondary Outcome: Proportion of Subjects Achieving 75% Reduction at Each Visit
Description: Proportion of subjects achieving 75% reduction from baseline in number of molluscum contagiosum at each visit
Time Frame: Week 1, Week 2, Week 4, Week 8, Week 12
Population: mITT population.
Measure: Number; unit: participants
Arm/Group | Cohort 1: SB206 4% BID | Cohort 2: SB206 8% BID | Cohort 3: SB206 12% BID | Cohort 4: SB206 12% QD | Placebo (Vehicle Gel)
Number analyzed (Participants) | 38 | 39 | 37 | 43 | 60
participants
  Week 1 proportion of subjects achieving complete clearance.: number analyzed (Participants) | 35 | 37 | 36 | 43 | 57
  Week 1 proportion of subjects achieving complete clearance. | 1 | 1 | 3 | 3 | 1
  Week 2 proportion of subjects achieving complete clearance.: number analyzed (Participants) | 38 | 39 | 36 | 42 | 59
  Week 2 proportion of subjects achieving complete clearance. | 4 | 1 | 3 | 8 | 3
  Week 4 proportion of subjects achieving complete clearance.: number analyzed (Participants) | 37 | 39 | 36 | 41 | 59
  Week 4 proportion of subjects achieving complete clearance. | 4 | 6 | 9 | 9 | 5
  Week 8 proportion of subjects achieving complete clearance.: number analyzed (Participants) | 37 | 37 | 36 | 41 | 58
  Week 8 proportion of subjects achieving complete clearance. | 8 | 14 | 18 | 20 | 11
  Week 12 proportion of subjects achieving complete clearance.: number analyzed (Participants) | 34 | 39 | 36 | 43 | 59
  Week 12 proportion of subjects achieving complete clearance. | 10 | 20 | 20 | 22 | 18

5. Secondary Outcome: Mean Change in Molluscum Contagiosum at Each Visit
Description: Mean change from baseline in number of molluscum contagiosum lesions at each visit
Time Frame: Week 1, Week 2, Week 4, Week 8, Week 12
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: Molluscum lesion counts
Arm/Group | Cohort 1: SB206 4% BID | Cohort 2: SB206 8% BID | Cohort 3: SB206 12% BID | Cohort 4: SB206 12% QD | Placebo (Vehicle Gel)
Number analyzed (Participants) | 38 | 39 | 37 | 43 | 60
Molluscum lesion counts
  Week 1: number analyzed (Participants) | 35 | 37 | 36 | 43 | 57
  Week 1 | -1.5 (1.43) | 0 (1.33) | -2.5 (1.44) | -4.0 (1.27) | 0.7 (1.13)
  Week 2: number analyzed (Participants) | 38 | 39 | 36 | 42 | 59
  Week 2 | -1.9 (1.53) | -1.7 (1.45) | -1.8 (1.57) | -7.1 (1.41) | -1.2 (1.23)
  Week 4: number analyzed (Participants) | 37 | 39 | 36 | 41 | 59
  Week 4 | -1.8 (1.80) | -6.0 (1.71) | -6.2 (1.82) | -8.7 (1.66) | -0.9 (1.43)
  Week 8: number analyzed (Participants) | 37 | 37 | 36 | 41 | 58
  Week 8 | -5.6 (2.08) | -10.3 (2.00) | -7.6 (2.10) | -12.3 (1.92) | -4.9 (1.65)
  Week 12: number analyzed (Participants) | 34 | 39 | 36 | 43 | 59
  Week 12 | -7.2 (2.43) | -12.0 (2.31) | -9.9 (2.42) | -12.9 (2.21) | -8.6 (1.90)

6. Secondary Outcome: Percent Change in Molluscum Contagiosum at Each Visit
Description: Percent change from baseline in number of molluscum contagiosum lesions at each visit
Time Frame: Week 1, Week 2, Week 4, Week 8, Week 12
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | Cohort 1: SB206 4% BID | Cohort 2: SB206 8% BID | Cohort 3: SB206 12% BID | Cohort 4: SB206 12% QD | Placebo (Vehicle Gel)
Number analyzed (Participants) | 38 | 39 | 37 | 43 | 60
Percentage change from baseline
  Week 1: number analyzed (Participants) | 35 | 37 | 36 | 43 | 57
  Week 1 | 0.0 (7.82) | 10.1 (7.33) | -4.7 (7.84) | -11.1 (6.96) | 8.7 (6.16)
  Week 2: number analyzed (Participants) | 38 | 39 | 36 | 42 | 59
  Week 2 | -4.4 (8.44) | 5.8 (8.07) | -5.9 (8.64) | -29.2 (7.81) | -4.1 (6.77)
  Week 4: number analyzed (Participants) | 37 | 39 | 36 | 41 | 59
  Week 4 | -3.6 (8.19) | -30.4 (7.75) | -29.2 (8.32) | -37.3 (7.54) | -6.6 (6.51)
  Week 8: number analyzed (Participants) | 37 | 37 | 36 | 41 | 58
  Week 8 | -19.2 (9.54) | -47.5 (9.17) | -38.7 (9.64) | -56.3 (8.79) | -17.2 (7.58)
  Week 12: number analyzed (Participants) | 34 | 39 | 36 | 43 | 59
  Week 12 | -25.3 (9.65) | -64.3 (9.07) | -56.1 (9.61) | -54.6 (8.70) | -37.8 (7.54)

ADVERSE EVENTS:
Time Frame: Baseline visit to end of study visit, 85 days.
Description: The at risk population is based on the Safety Population. Only TEAEs were to be considered.
Groups:
- Cohort 3: SB206 12% BID: SB206 12%: topically twice daily
Arm/Group | Cohort 1: SB206 4% BID | Cohort 2: SB206 8% BID | Cohort 3: SB206 12% BID | Cohort 4: SB206 12% QD | Placebo (Vehicle Gel)
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/48 | 0/47 | 0/47 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48 | 0/47 | 0/47 | 0/66
Other Adverse Events (participants affected / at risk) | 7/46 | 24/48 | 18/47 | 19/47 | 6/66
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: SB206 4% BID (N=46) | Cohort 2: SB206 8% BID (N=48) | Cohort 3: SB206 12% BID (N=47) | Cohort 4: SB206 12% QD (N=47) | Placebo (Vehicle Gel) (N=66)
Application site erythema (General disorders) | 3 | 6 | 6 | 5 | 0
Application site pain (General disorders) | 2 | 3 | 3 | 4 | 0
Pyrexia (General disorders) | 1 | 5 | 1 | 1 | 2
Application site exfoliation (General disorders) | 0 | 1 | 3 | 4 | 0
Application site pruritus (General disorders) | 1 | 1 | 4 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 3 | 1 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must wait 18 months after the closeout of the trial at all Study sites or until the publication of the multi-site Sponsor results. The only restriction on PI publication after that time is that the sponsor can review results communications prior to public release and can request confidential or proprietary information be removed or can embargo communications regarding trial results for a period that is more than 90 days but less than 120 days.

DOCUMENTS (2):
  • Study Protocol (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT03436615/Prot_001.pdf
  • Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT03436615/SAP_002.pdf